CLINICAL TRIAL: NCT04317521
Title: A Prospective Study Investigating the Use of the Eko CORE and Eko DUO Electronic Stethoscopes for Differentiation of Innocent vs. Pathologic Murmurs in Pediatric Patients.
Brief Title: : A Prospective Study Investigating the Use of the Eko CORE and Eko DUO Electronic Stethoscopes in Pediatric Patients.
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1575863-1
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2021-01

CONDITIONS: Heart Murmurs
MeSH Terms: conditions — Heart Murmurs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Use of EKO Core and EKO Duo electronic stethoscopes — Listen to heart murmurs

SUMMARY:
The Eko CORE and DUO stethoscopes are FDA approved electronic devices which have the capacity to record heart sounds. This study will utilize these devices to see if they can differentiate between pathologic and innocent heart murmurs in children.

DETAILED DESCRIPTION:
It is estimated that 50-70% of all children will have had a detectable heart murmur at some point in early life, but fortunately, the vast majority of these murmurs are benign asymptomatic "innocent" murmurs and not indicative of heart disease. However, there is concern about the ability of front-line pediatricians and family providers to distinguish between an innocent and pathological murmur. Thus, it is of no surprise that the largest number of new patient referrals to pediatric cardiologists is due to the detection of a murmur. Of those referred, 20-30% are typically diagnosed with trivial to significant heart disease based on auscultation and confirmatory echocardiography follow-up when necessary.

Having a child referred for a heart murmur evaluation causes significant anxiety for parents, even if the murmur is suggested to be innocent by the pediatrician and in some cases, clinical diagnostic testing is done unnecessarily. Interestingly, studies have shown that performing diagnostic electrocardiography, chest radiography, or echocardiography prior to clinical assessment by pediatric cardiologists did not offer additional assistance in differentiating murmurs. Unnecessary echocardiograms or other diagnostic tests for innocent murmur evaluation add unnecessary cost to the healthcare system.

Unfortunately, the unnecessary use of echocardiography for the diagnosis of innocent murmurs is also high among pediatric cardiologists. Thus, with the rising cost of health care, it is essential that we identify and target areas of practice that will enable us to increase efficiency and reduce unnecessary costs.

Specific characteristics of the sound of the murmur may help differentiate innocent from other murmurs, so improving auscultation skills and diagnosis based on auscultation and electrocardiography is very important in accurate diagnosis and reducing cost associated with the diagnosis of innocent and pathologic heart murmurs in children. The use of new technologies to improve auscultation and auscultation-based diagnosis could lead to improved diagnoses with decreased cost. New systems that used telemedicine techniques to transfer phonocardiogram (PCG) recordings to a cloud server have shown benefit in differentiating innocent versus pathologic murmurs, but cannot be used large scale, and are based on cardiology involvement.

The FDA-cleared Eko CORE device (Eko, Berkeley, California, USA) is a digital stethoscope that allows recording of the audio to produce a PCG. The FDA-cleared Eko DUO device is a digital stethoscope that allows recording of the audio to produce a PCG combined with a single lead electrocardiograph. The CORE and DUO both feature sound amplification and audio transmission to a smart phone, laptop or tablet via Bluetooth® that allows the user to open and playback sounds using an iOS, Android, or Microsoft Windows compatible application. The App provides the ability to save sounds within select Electronic Health Record (EHR) systems, share patient recordings with other practitioners, and annotate notes on recorded audio. Eko is intended for use on pediatric and adult patients. These features uniquely situate this device to accumulate large sets of auscultatory data on patients both with and without congenital heart disease (CHD).

In this study, we seek to use auscultatory audio recordings and phonocardiograms collected from pediatric patients using Eko CORE and DUO digital stethoscopes to develop a clinically significant algorithm that differentiates innocent from pathologic heart murmurs. As the Eko CORE and DUO devices are similar to a traditional stethoscope, an iconic tool widely accepted by patients and providers alike, its use to drive an automated detection algorithm is both feasible and attractive as a substitute for traditional auscultation. Furthermore, by providing an algorithmic analysis that can supplement clinical acumen, we hypothesize that we will improve overall diagnostic accuracy and show a decreased need for referral echocardiograms for innocent murmurs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 0 to 17 years, who are able to read and speak English, and/or with parents or legal guardians who are able to read and speak English
2. New patients referred to the Nemours Cardiac Center for a heart murmur, chest pain, syncope, or arrhythmia. This could include children with suspected murmurs (but ultimately found to have no murmur by a cardiologist), innocent murmurs, and pathologic murmurs.
3. Patients with previously diagnosed heart condition, if they have not had any corrective surgeries and had a detectable murmur at their last clinic visit (for pathological and innocent murmurs) or had no detectable murmur at their last clinic visit (for no murmurs).

Exclusion Criteria:

1. Patients aged 18 and over
2. Patients and/or parents who are unable to read or speak English
3. Patients who have had corrective heart surgery for a heart defect
4. Auscultation cannot be performed properly at all locations
5. Patients not wishing to participate in study recordings

Ages: 2 Days to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children attending the Nemours Cardiac Center to include patients referred for a heart murmur who are aged from 0 to 17 years, patients with previously diagnosed heart conditions, patent ductus arteriosus (PDA) or valvular stenosis, who have not undergone corrective surgery and had a detectable murmur at their last visit. Patients who have an innocent or no detectable heart murmur will be from new referrals for a heart murmur, chest pain, syncope, or arrhythmia, or are currently outpatients in the cardiac clinic who had an innocent murmur or no detectable heart murmur in their previous (and current) clinic appointments, and meet the inclusion/exclusion criteria for the study.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Comparison of stethoscope recordings between innocent, pathologic and none to determine if stethoscope can differentiate | Recording 2 minutes of heart sounds for each stethoscope
  The data science team will generate ROC curves for algorithm scores in the set of recorded heart sounds. Exploratory descriptive analyses of the algorithm will be performed by identifying clinical correlates to the characteristics most heavily weighted in detecting a pathologic murmur. The likelihood ratios of the test at sensitivity cut offs of 0.90, 0.95, 0.99 will also be determined.
  Patients will also be stratified based on age as a secondary outcome: For example, infants (0<1 years of age, since murmurs in this age group are more likely to be pathologic), young children (1-5 years of age), children (>5-12 years of age) and adolescents (>12 to<18 years of age). Murmurs will be classified as none, innocent [defined as no significant heart disease on echocardiogram and further classified as Still's, pulmonary flow murmur, systemic flow murmur, venous hums by the physician], or pathological by disease type (e.g., atrial septal defect (ASD), ventricular septal defect (VSD), etc.

SECONDARY OUTCOMES:
Murmurs identified by stethoscope recording will be stratified based on age | 2 minutes of recording with two stethoscopes
  Differentiated murmurs of infants between 0-1 years, young children, ages 1-5 years, children ages >5-12 years and adolescents >12 years < 18 years will be evaluated and murmurs identified

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Slamon, MD, Principal Investigator — Nemours/Alfred I duPont Hospital for Children
Locations (1):
- Nemours Alfred I duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose-Felker K, Kelleman MS, Campbell RM, Oster ME, Sachdeva R. Appropriate Use and Clinical Impact of Echocardiographic "Evaluation of Murmur" in Pediatric Patients. Congenit Heart Dis. 2016 Dec;11(6):721-726. doi: 10.1111/chd.12379. Epub 2016 Jun 10. PMID 27282847
- [Background] Sachdeva R, Allen J, Benavidez OJ, Campbell RM, Douglas PS, Eidem BW, Gold L, Kelleman MS, Lopez L, McCracken CE, Stern KW, Weiner RB, Welch E, Lai WW. Pediatric Appropriate Use Criteria Implementation Project: A Multicenter Outpatient Echocardiography Quality Initiative. J Am Coll Cardiol. 2015 Sep 8;66(10):1132-40. doi: 10.1016/j.jacc.2015.06.1327. PMID 26337992
- [Background] Rose-Felker K, Kelleman MS, Campbell RM, Sachdeva R. Appropriateness of Outpatient Echocardiograms Ordered by Pediatric Cardiologists or Other Clinicians. J Pediatr. 2017 May;184:137-142. doi: 10.1016/j.jpeds.2017.01.073. Epub 2017 Feb 24. PMID 28238480
- [Background] Kourtidou S, Evers PD, Jorgensen NW, Kronmal RA, Lewin MB, Schultz AH. Pediatric Appropriate Use Criteria for Outpatient Echocardiography: Practice Variations among Pediatric Cardiologists, Noncardiologist Subspecialists, and Primary Care Providers. J Am Soc Echocardiogr. 2017 Dec;30(12):1214-1224. doi: 10.1016/j.echo.2017.08.014. Epub 2017 Nov 1. PMID 29079043
- [Background] Yi MS, Kimball TR, Tsevat J, Mrus JM, Kotagal UR. Evaluation of heart murmurs in children: cost-effectiveness and practical implications. J Pediatr. 2002 Oct;141(4):504-11. doi: 10.1067/mpd.2002.127502. PMID 12378189
- [Background] Pyles L, Hemmati P, Pan J, Yu X, Liu K, Wang J, Tsakistos A, Zheleva B, Shao W, Ni Q. Initial Field Test of a Cloud-Based Cardiac Auscultation System to Determine Murmur Etiology in Rural China. Pediatr Cardiol. 2017 Apr;38(4):656-662. doi: 10.1007/s00246-016-1563-8. Epub 2017 Feb 2. PMID 28150025
- [Background] Gardezi SKM, Myerson SG, Chambers J, Coffey S, d'Arcy J, Hobbs FDR, Holt J, Kennedy A, Loudon M, Prendergast A, Prothero A, Wilson J, Prendergast BD. Cardiac auscultation poorly predicts the presence of valvular heart disease in asymptomatic primary care patients. Heart. 2018 Nov;104(22):1832-1835. doi: 10.1136/heartjnl-2018-313082. Epub 2018 May 24. PMID 29794244
- [Background] Chambers J, Kabir S, Cajeat E. Detection of heart disease by open access echocardiography: a retrospective analysis of general practice referrals. Br J Gen Pract. 2014 Feb;64(619):e105-11. doi: 10.3399/bjgp14X677167. PMID 24567615
- [Background] Danford DA, Nasir A, Gumbiner C. Cost assessment of the evaluation of heart murmurs in children. Pediatrics. 1993 Feb;91(2):365-8. PMID 8424012
- [Background] McCrindle BW, Shaffer KM, Kan JS, Zahka KG, Rowe SA, Kidd L. Cardinal clinical signs in the differentiation of heart murmurs in children. Arch Pediatr Adolesc Med. 1996 Feb;150(2):169-74. doi: 10.1001/archpedi.1996.02170270051007. PMID 8556121
- [Background] Mackie AS, Jutras LC, Dancea AB, Rohlicek CV, Platt R, Beland MJ. Can cardiologists distinguish innocent from pathologic murmurs in neonates? J Pediatr. 2009 Jan;154(1):50-54.e1. doi: 10.1016/j.jpeds.2008.06.017. Epub 2008 Aug 9. PMID 18692204
- [Background] Draper J, Subbiah S, Bailey R, Chambers JB. Murmur clinic: validation of a new model for detecting heart valve disease. Heart. 2019 Jan;105(1):56-59. doi: 10.1136/heartjnl-2018-313393. Epub 2018 Jul 26. PMID 30049836
- [Background] Frias PA, Oster M, Daley PA, Boris JR. Outpatient echocardiography in the evaluation of innocent murmurs in children: utilisation benchmarking. Cardiol Young. 2016 Mar;26(3):499-505. doi: 10.1017/S1047951115000517. Epub 2015 Apr 23. PMID 25902744
- [Background] Hajian-Tilaki K. Sample size estimation in diagnostic test studies of biomedical informatics. J Biomed Inform. 2014 Apr;48:193-204. doi: 10.1016/j.jbi.2014.02.013. Epub 2014 Feb 26. PMID 24582925
- See also: website for FDA approved devices — http://www.ekohealth.com